CLINICAL TRIAL: NCT02781233
Title: The Impact of Progressive Resistance Training on Quality of Life in Patients With Haemophilia
Brief Title: A Progressive Resistance Training Program in Patients With Haemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Felipe Querol Fuentes, Medical doctor, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H15-29504
Record Dates: First submitted 2016-05-18; First posted 2016-05-24 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Each subject will participate in 2 sessions each week during 8 weeks, with 3 days of difference (rest) between the sessions.
  Interventions: Other: Progressive resistance training
- Control group (Placebo Comparator): Usual daily activities
  Interventions: Other: Normal daily activities

INTERVENTIONS:
Other: Progressive resistance training — Progressive resistance training program
  Arms: Training group
Other: Normal daily activities — Usual daily activities
  Arms: Control group

SUMMARY:
This study evaluates the clinical impact of a progressive resistance training program in adults patients with haemophilia

DETAILED DESCRIPTION:
The training program aims improving muscular strength and endurance in the relevant muscles and joints (knee, elbow, ankle, shoulder and hip) in order to improve the quality of life in the patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of haemophilia A or B
* willingness to exercise twice a week during the training program and to complete the pre- and post-program evaluations
* approval by their hematologist to participate in the exercise program
* age between 18 and 60 years
* informed consent signed.

Exclusion Criteria:

* the inability to attend exercise sessions at least twice a week for 6 consecutive weeks
* non adherence to instruction on proper exercise technique
* surgical procedures performed 6 weeks prior to or during the exercise program
* participation in any other form of exercise, including rehabilitation, during the study; (5) changes in medication during the study
* a major bleeding episode that posed a risk or prevented exercise
* History of FVIII inhibitor (titer ≥ 0.6 BU [Bethesda unit]) or detectable FVIII inhibitors at screening (titer ≥ 0.4 BU)
* Another haemostatic defect
* Need for major surgery
* Withdrawal of informed consent

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Change in Muscle strength | baseline and 8 weeks
  For measuring the isometric knee flexion and extension, ankle plantarflexion and dorsiflexion strength and isometric elbow flexion and extension strength, a portable hand-held dynamometer will be used (Nicholas Manual Muscle Tester, Lafayette Instruments, Indiana, USA).

SECONDARY OUTCOMES:
Change in Timed Up and Go | baseline and 8 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Change in Haemophilia Quality of life questionnaire (A36 Haemophilia-QoL® ) | baseline and 8 weeks
  The Haemophilia-QoL questionnaire is a self-report modular instrument that assesses nine relevant HRQoL domains for patients with haemophilia (e.g. physical health, daily activities, joint damage, pain, treatment satisfaction, treatment difficulties, emotional functioning, mental health, relationships and social activity).
Change in Bleedings | daily (during the 8 weeks of intervention)
  Number of Bleedings During the study
Change in viscoelastic properties (rectus femoris) | baseline and 8 weeks
  Myoton Pro
Change in sit-to-stand test | baseline and 8 weeks
  The time taken for the participant to stand up and sit down from a standard 45 cm chair with arms three times, as quickly as possible, was measured.
Change in Haemophilia Activities List questionnaire | baseline and 8 weeks
  The Haemophilia Activities List questionnaire measures the impact of hemophilia on self-perceived functional abilities in adults.
  It contains 42 multiple choice questions in seven domains:
  Lying/sitting/kneeling/standing (8 items) Functions of the legs (9 items) Functions of the arms (4 items) Use of transportation (3 items) Self-care (5 items) Household tasks (6 items) Leisure activities and sports (7 items) The most important outcomes are the overall sum score and three component scores relating to upper extremity activities, basic lower extremity activities, and complex lower extremity activities. A domain score for each of the seven domains can also be calculated.
Change in The Haemophilia Joint Health Score (HJHS) | baseline and 8 weeks
  The HJHS measures joint health, in the domain of body structure and function (i.e. impairment), of the joints most commonly affected by bleeding in hemophilia: the knees, ankles, and elbows.The HJHS 2.1 provides a total score (higher score is worse; max=124), joint specific scores, and a global gait score.
Change in Pain | baseline and 8 weeks
  11-point numerical pain rating scale with higher score meaning higher pain
Change in workability index | baseline and 8 weeks
  workability index with single question
Change in analgesics use (days/week) | baseline and 8 weeks
  The number of days the participants used analgesics during the last week
Change in Range Of Motion (ROM) | baseline and 8 weeks
  elbow extensio/flexion, ankle dorsiflexion/plantar flexion and knee flexion/extension ROM with a goniometer
Change in Kinesiophobia | baseline and 8 weeks
  Tampa Scale of Kinesiophobia (TSK-11SV) used to assess changes in fear of movement

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Querol-Fuentes, MD, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calatayud J, Perez-Alenda S, Carrasco JJ, Cruz-Montecinos C, Andersen LL, Bonanad S, Querol F, Megias-Vericat JE, Casana J. Safety and Effectiveness of Progressive Moderate-to-Vigorous Intensity Elastic Resistance Training on Physical Function and Pain in People With Hemophilia. Phys Ther. 2020 Aug 31;100(9):1632-1644. doi: 10.1093/ptj/pzaa106. PMID 32525975